CLINICAL TRIAL: NCT02386410
Title: Selective Prevention of Anxiety Disorders in Children: A Randomized Controlled Preliminary Study of a Parent Training Intervention for Anxious Parents
Brief Title: Selective Prevention of Anxiety Disorders in Children: A Parent Training Intervention for Anxious Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ata Ghaderi, Professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AGJA-02
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group parent training (Experimental): The intervention Group parent training for anxious parents is delivered in groups of about five, in 90 minutes per session, for eight consecutive weeks. The parent training is delivered by a licensed psychologist.
  Interventions: Behavioral: Group parent training for anxious parents
- Internet delivered parent training (Experimental): In the internet delivered parent training for anxious parents, parents are asked to work with one chapter each week, for eight consecutive weeks. Each chapter mirrors a session in the group format. Parents are able to e-mail a licensed psychologist during the intervention.
  Interventions: Behavioral: Internet delivered parent training for anxious parents
- Wait-list (No Intervention): Parents in the wait-list condition will receive the intervention after 12-month follow-up.

INTERVENTIONS:
Behavioral: Group parent training for anxious parents
  Arms: Group parent training
Behavioral: Internet delivered parent training for anxious parents
  Arms: Internet delivered parent training

SUMMARY:
Anxiety is the most frequent psychiatric problem in children. Untreated anxiety often has a chronic course, or may be a recurring condition. Anxiety in children predicts a variety of psychiatric disorders later in life, and involves problems regarding school performance and social relations. The literature provides a number of factors, which are suggested to increase the risk of developing an anxiety disorder. In particular, it has been shown that children of parents with anxiety disorders are at much greater risk of developing an anxiety disorder. Several studies have found a correlation between anxiety in the child, and parent behavior characterized by criticism, control and overprotectiveness. The present study aim to preliminary evaluate whether a eight week parent training intervention can reduce the incidence of anxiety disorders in children and to evaluate the feasibility of the parent training. Three central factors has been the basis in developing the parent training, all of which are considered to be involved in the development and maintenance of anxiety disorders in children (1) criticism and rejection, (2) control and overprotectiveness, and (3) parental modeling and reinforcement of anxiety. The goal of the parent training is therefore (1) to increase warmth and acceptance, (2) to increase autonomy for the child, and (3) modeling and reinforcement of brave behavior. The investigators intend to include 60 anxious parents in the study, who will be randomly allocated to either group parent training, Internet delivered parent training, or wait-list condition. The inclusion criteria are as follows: The parent states that he/she experiences anxiety or worry, the parents' child is 6-12 years old, and do not fulfill criteria for an anxiety disorder or major depressive disorder, the parent possesses everyday access to the Internet, and there is no presence of very aggravated family situations, such as parent substance abuse or severe depression, or domestic violence.

ELIGIBILITY:
Inclusion Criteria:

* The parent states that he/she experiences anxiety or worry,
* The parents' child is 6-12 years old, and do not fulfill criteria for an anxiety disorder or major depressive disorder
* The parent possesses everyday access to the Internet

Exclusion Criteria:

* Presence of very aggravated family situations, such as parent substance abuse or severe depression, or domestic violence.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule - Child and Parent Version | At 12-month follow up

SECONDARY OUTCOMES:
The Spence Children's Anxiety Scale | Change from baseline in anxiety symptom scores at 12 months follow-up
  Rated by the child and the parent independently
Children Depression Inventory | Change from baseline in depressive symptom scores at 12 months follow-up
  Rated by the child
The Rearing Behavior Questionnaire | Change from baseline in rearing behavior scores at 12 months follow-up
  Rated by parents
Strengths and Difficulties Questionnaire | Change from baseline in dfficulties scores at 12 months follow-up
  Rated by parents
State-Trait Anxiety Inventory | Change from baseline in anxiety symptom scores at 12 months follow-up
  Rated by parents
Montgomery-Åsberg Depression Rating Scale | Change from baseline in depressive symptom scores at 12 months follow-up
  Rated by parents
Quality of Life Inventory | Change from baseline in quality of life scores at 12 months follow-up
  Rated by parents

CONTACTS AND LOCATIONS:
Overall Officials: Ata Ghaderi, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden